CLINICAL TRIAL: NCT03946683
Title: Cyberknife Radiosurgery for Early Stage Breast Cancer: A Winthrop-University Hospital Pilot Study of Cyberknife Partial Breast Radiosurgery for Tumors 3 cm or Less
Brief Title: Cyberknife for Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-01721; 18-01721 (Other: NYU Langone Institutional Review Board)
Record Dates: First submitted 2015-01-05; First posted 2019-05-13 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Early Stage Breast Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyberknife for Early Stage Breast Cancer (Experimental): Cyberknife Robotic Radiosurgery will be utilized as a 5-fraction post-lumpectomy adjuvant radiation treatment in the management of early stage breast cancer.
  Interventions: Radiation: Cyberknife for Early Stage Breast Cancer

INTERVENTIONS:
Radiation: Cyberknife for Early Stage Breast Cancer — Utilization of Cyberknife Robotic Radiosurgery as a 5-fraction post-lumpectomy adjuvant radiation treatment in the management of early stage breast cancer
  Other Names: SBRT (Stereotactic Body Radiation Therapy)

SUMMARY:
This phase II study based on the Cyberknife Society study will evaluate the technical feasibility and acute toxicity of Partial Breast Irradiation (PBI) with the Cyberknife. It will evaluate quality of life (QOL) issues as they relate to treatment-related side effects, cosmetic result and patient convenience. It will evaluate outcome in terms of local control in the treated breast.

Radiosurgery is defined as the stereotactic delivery of ionizing radiation in 5 stages or less to a designated target with sub-millimeter accuracy. Radiosurgery in the context of this protocol will be given to the region of the tumor bed with 7 weeks of the lumpectomy and sent/axillary node sampling over the period of five to ten days using the Cyberknife (CK) or within the 7 weeks of the last chemotherapy treatment if given.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 0, I, or II (Tis, Ti, or T2 <=3cm & NO) histologically confirmed invasive non-lobular carcinoma or ductal carcinoma in situ of the breast with a lesion <= 3 cm, treated with wide excision.
* Negative inked histologic margins of excision or reexcision and clear of invasive tumor and DClS by at least 2mm
* Negative post-excision or post-reexcision mammography if cancer presented with malignancy-associated microcalcifications; no remaining suspicious microcalcifications in the breast before radiotherapy.
* No involved axillary lymph nodes by routine histologic examination (H&E) of sentinel node(s) or of nodes identified from axillary dissection.
* Enrollment and initiation of CyberKnife therapy within 42 days of last breast cancer surgery or last chemotherapy treatment.

Exclusion Criteria:

* Patients with invasive lobular carcinoma or nonepithelial breast malignancies such as sarcoma or lymphoma.
* Patients with multicentric carcinoma or with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy.
* Patients who are pregnant.
* Patients who have any histologically confirmed positive axillary nodes.
* Patients with collagen vascular diseases, specifically systemic lupus erythematosis, scleroderma, or dermatomyositis with a creatine phosphokinase level above normal or with an active skin rash.

Ages: 45 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Local Control Rate | 1 Year
  Mastectomy-free survival rate after Cyberknife body radiosurgery [Mastectomy and death will be considered failures]

SECONDARY OUTCOMES:
Complication Rate | 1 Year
  Rate of complications or toxicities after Cyberknife body radiosurgery (including skin reactions to radiotherapy and any acute complications or unusual side effects) will be measured via physician's observation and via toxicity reports.
Score on The Harvard/NSABP/RTOG Breast Cosmesis Scale. | Baseline, week 10, and week 26
  4 Point Scale (I-IV): I. Excellent: When compared with the untreated breast, there is minimal or no difference in the size or shape of the treated breast. II. Good: There is a slight difference in the size or shape of the treated breast as compared with the opposite breast or the original appearance of the treated breast. There may be some mild reddening or darkening of the breast. The thickening or scar tissue III. Fair: Obvious difference in the size and shape of the treated breast. This change involves one-quarter or less of the breast. IV. Poor: Marked change in the appearance of the treated breast involving more than onequarter of the breast tissue. The skin changes may be obvious and detract from the appearance of the breast.
Measure of self reported quality of life using the QOLS | 1 Year
  41-item survey can be administered by interviewed in person or over the telephone, and it may also be self-administered by respondents with adequate cognitive functioning. The questions are divided into 5 categories-Material and Physical Well-being, Relationships with other People, Social, Community, and Civic Activities, Personal Development and Fulfillment and Recreation.The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A. Haas, MD, Principal Investigator — NYU Winthrop Hospital
Locations (1):
- NYU Langone Health, New York, New York, United States

REFERENCES:
- See also: CyberKnife Radiosurgery for Early-Stage Breast Cancer — http://www.disabled-world.com/medical/surgery/cyberknife-radiosurgery.php
- See also: University of Texas Southwestern launches clinical trial for treatment of breast cancer using robotic CyberKnife technology — http://www.utsouthwestern.edu/utsw/cda/dept353744/files/628373.html